CLINICAL TRIAL: NCT02908178
Title: Comparative Effectiveness of Sentinel Lymph Node Biopsy (SLNB) for Ductal Carcinoma In Situ (DCIS)
Brief Title: Comparative Effectiveness of Sentinel Lymph Node Biopsy for Ductal Carcinoma In Situ
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI-SW-1
Record Dates: First submitted 2016-08-30; First posted 2016-09-20 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Ductal Carcinoma In Situ
Keywords: ductal carcinoma in situ (DCIS); sentinel lymph node biopsy (SLNB)
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aim 1 Cohort: The Aim 1 Cohort is constructed to perform analysis to address study objective Aim 1. This cohort includes patients diagnosed at ages 67-94 years with DCIS between January 1998 and December 2011, and received BCS as their first surgery. Patients in this cohort include those who received sentinel lymph node biopsy (SLNB) and who didn't receive SLNB.
  The Aim 1 Cohort and the Aim 2 Cohort can overlap.
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB)
- Aim 2 Cohort: The Aim 2 Cohort is constructed to perform analysis to address study objective Aim 2. This cohort includes patients diagnosed at ages 67-94 years with DCIS between January 2001 and December 2013, and received BCS as their first surgery. Patients in this cohort include those who received sentinel lymph node biopsy (SLNB) and who didn't receive SLNB.
  The Aim 1 Cohort and the Aim 2 Cohort can overlap.
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB)

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy (SLNB) — Intervention is defined as that the DCIS patient has undergone SLNB. Patients in each cohort (group) include those who underwent SLNB (intervention) and those who did not (control).

SUMMARY:
Patients with ductal carcinoma in situ (DCIS) treated with available therapies have experienced excellent outcomes and very low mortality rates due to the disease's non-invasive nature. However, considerable debate exists as to how the DCIS lesion should be treated. As a result, determining strategies to manage DCIS has been identified as a research priority. The role of sentinel lymph node biopsy (SLNB) for DCIS management is controversial in general and needs further scrutiny. Our study addresses this evidence gap as the investigators propose a retrospective cohort study to investigate the outcome of SLNB among DCIS patients. Specifically, the investigators will compare the outcomes, including survival outcomes and treatment side effects, among women older than 67 years of age with DCIS receiving SLNB vs. not receiving SLNB within 6 months of DCIS diagnosis. The investigators have two primary aims in this study: Aim 1: the investigators select our study sample using SEER-Medicare database. The investigators will determine associations between SLNB and acute/subacute side effects, including lymphedema, pain, and limitation of movement of upper extremity from the first breast conserving surgery to 9 months post-diagnosis. Aim 2: the investigators will determine associations between SLNB and long-term outcomes, including breast cancer specific mortality, ipsilateral invasive breast cancer diagnosis, subsequent mastectomy as treated recurrence, and lasting side effects, from >9 months post-diagnosis to death or the end of this study period.

Given the nature of our observational study design, the investigators will apply standard multivariate analyses and propensity score methodology to reduce the influence from confounders. The investigators will control for patient demographics, comorbidities, functional status, tumor characteristics, and prior healthcare utilization. Using distance to the nearest provider that uses SLNB for DCIS or surgeon's tendency in using SLNB for stage I/II breast cancer, the investigators also plan to conduct instrument variable analyses if necessary. Stratifying patients by key DCIS characteristics (including grade, comedonecrosis, and tumor size) and their predicted life expectancy (given their age and comorbidities), the investigators also hope to identify patient subgroups who may safely forgo SLNB. The study would provide evidence on the efficacy and safety outcome of SLNB for DCIS management.

DETAILED DESCRIPTION:
Because of the non-invasive nature of ductal carcinoma in situ (DCIS), patients treated with available therapies have excellent outcomes and very low rates of breast cancer mortality. Considerable debate exists as to how the DCIS lesion should be treated, although there is a movement toward less intensive intervention by the identification of patient subsets with favorable prognoses. Some prospective studies have found that the rate of ipsilateral invasive cancer occurrence is still high after receiving breast conserving surgery (BCS) alone, even among patients with favorable pathologic characteristics. Such findings argue against active surveillance for DCIS treatment. However, evidence exists that older DCIS patients have a lower rate of ipsilateral recurrence because DCIS among older patients tends to be indolent. Identifying suitable subgroups among this lower risk group who may be safe to receive a less aggressive treatment could change the current practice pattern of aggressive treatment.

Even when DCIS patients opt to receive a less intensive treatment such as BCS without radiation therapy, they and their providers need to decide whether to undergo sentinel lymph node biopsy (SLNB). A systematic review has shown that evidence gaps exist regarding the benefits of SLNB for DCIS. Given that the likelihood of axillary recurrence is low among DCIS patients who received radiation therapy, routine SLNB is not recommended for DCIS patients. Of note, radiation therapy can control axillary disease if present. If the investigators plan to empower DCIS patients to choose less intensive management options, such as BCS forgoing radiation therapy (RT), it will be crucial for patients and providers to understand the role of SLNB.

The overarching goals of this study are to compare side effects and outcomes between receiving SLNB vs. not receiving SLNB among older DCIS patients who received BCS. With this data, the investigators also aim to identify sub-populations for whom less intensive treatments may be appropriate. Using the Surveillance, Epidemiology, and End Result (SEER)-Medicare linked data, our project's overarching aims are:

Among older women with DCIS who have received BCS as their first surgery, to compare the outcomes of receiving sentinel lymph node biopsy (SLNB) vs. not receiving SLNB within 6 months of DCIS diagnosis:

Aim 1: The investigators will determine associations between SLNB and acute/subacute side effects, including lymphedema, pain, and limitation of movement of upper extremity from the first BCS to 9 months post-diagnosis Aim 2: The investigators will determine associations between SLNB and long-term outcomes, including breast cancer specific mortality, ipsilateral invasive breast cancer diagnosis, subsequent mastectomy as treated recurrence, and lasting side effects, from > 9 months' post-diagnosis to death or the end of the study period.

Our study is a retrospective cohort study with the study population being DCIS patients older than 67 years (hereafter referred to as older women) who were enrolled in a fee-for-service Medicare program and resided in the SEER areas from 1998 to 2011 (2001 to 2013 for Aim 2) and who were followed up to 2012 (2015 for Aim 2). The investigators selected age 67 years as a cut-off value because the investigators plan to use two years of claims data to identify patient comorbidities and control for them in our statistical models, and data is first available at age 65. Given the nature of our observational study design, the investigators will apply standard multivariate analyses and propensity score methodology to reduce the influence from confounders. The investigators will control for patient demographics, comorbidities, functional status, tumor characteristics, and prior healthcare utilization. Using distance to the nearest provider that uses SLNB for DCIS or surgeon's tendency in using SLNB for stage I/II breast cancer, the investigators also plan to conduct instrument variable analyses if necessary. Stratifying patients by key DCIS characteristics (including grade, comedonecrosis, and tumor size) and their predicted life expectancy (given their age and comorbidities), the investigators also hope to identify patient subgroups who may safely forgo SLNB.

In comparisons of baseline characteristics between intervention and control groups, the investigators will conduct standard descriptive statistics using chi-square tests for categorical variables and t-tests for continuous variables. The investigators will tabulate the frequencies of outcomes of interests by the intervention vs. control group. For multivariable analyses, the investigators will apply proportional hazards models to test whether the intervention is associated with better outcomes.

the investigators plan to control for this issue using propensity score matching methodology. Prior literature has suggested inclusion of either all measured variables or those variables that are associated with treatment selection (SLNB status) when conducting an analysis using the propensity score method. Specifically, our approach to matching will be based on the Mahalanobis distance calculated using age, race, residence in a metropolitan county, comorbidity, prior influenza vaccination or prior visit to a primary care physician (both as proxies for access to care), income, preoperative MRI use, and tumor characteristics. Tumor characteristics include size, grade, comedonecrosis, and estrogen receptor status. By incorporating these factors in matching, the investigators expect to substantially decrease bias and balance the risk for outcomes of interest between the SLNB and non-SLNB groups. The difference in outcomes between the control and intervention groups will be estimated in a Kaplan-Meier curve. The investigators will estimate the relative risk in the propensity score matched sample using the standard method for matched-pair data. The investigators will use the Cox proportional hazards models to investigate the association between various factors (grade, tumor size, and estrogen receptor status) and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female DCIS patients older than 67 years and younger than 94 years who were enrolled in a fee-for-service Medicare program and resided in the SEER areas.
* Aim 1: DCIS patients who received breast conserving surgery (BCS) as their first surgery
* Aim 1: DCIS patients who were diagnosed DCIS between January 1998 and December 2011
* Aim 2: DCIS patients who were diagnosed DCIS between January 2001 and December 2013

Exclusion Criteria:

* Aim 1: DCIS patients who received mastectomy as their first surgery
* Aim 2: DCIS patients who received BCS at the beginning yet received mastectomy in the end

Ages: 67 Years to 94 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Our study populations were generated within the SEER-Medicare linked database. The populations consist of female DCIS patients ages 67-94 years who were enrolled in a fee-for-service Medicare program and resided in the SEER areas.
Sampling Method: Non-Probability Sample
Enrollment: 28291 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Yi Wang, MD, PhD, Principal Investigator — Yale University
Locations (1):
- SEER-Medicare Dataset, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burstein HJ, Polyak K, Wong JS, Lester SC, Kaelin CM. Ductal carcinoma in situ of the breast. N Engl J Med. 2004 Apr 1;350(14):1430-41. doi: 10.1056/NEJMra031301. No abstract available. PMID 15070793
- [Background] American Cancer Society. Cancer Facts & Figure 2013. Atlanta: American Cancer Soc; 2013
- [Background] Virnig BA, Wang SY, Shamilyan T, Kane RL, Tuttle TM. Ductal carcinoma in situ: risk factors and impact of screening. J Natl Cancer Inst Monogr. 2010;2010(41):113-6. doi: 10.1093/jncimonographs/lgq024. PMID 20956813
- [Background] Allegra CJ, Aberle DR, Ganschow P, Hahn SM, Lee CN, Millon-Underwood S, Pike MC, Reed SD, Saftlas AF, Scarvalone SA, Schwartz AM, Slomski C, Yothers G, Zon R. National Institutes of Health State-of-the-Science Conference statement: Diagnosis and Management of Ductal Carcinoma In Situ September 22-24, 2009. J Natl Cancer Inst. 2010 Feb 3;102(3):161-9. doi: 10.1093/jnci/djp485. Epub 2010 Jan 13. PMID 20071686
- [Background] Gierisch JM, Myers ER, Schmit KM, Crowley MJ, McCrory DC, Chatterjee R, Coeytaux RR, Kendrick A, Sanders GD. Prioritization of research addressing management strategies for ductal carcinoma in situ. Ann Intern Med. 2014 Apr 1;160(7):484-91. doi: 10.7326/M13-2548. PMID 24567146
- [Background] Prendeville S, Ryan C, Feeley L, O'Connell F, Browne TJ, O'Sullivan MJ, Bennett MW. Sentinel lymph node biopsy is not warranted following a core needle biopsy diagnosis of ductal carcinoma in situ (DCIS) of the breast. Breast. 2015 Jun;24(3):197-200. doi: 10.1016/j.breast.2015.01.004. Epub 2015 Feb 11. PMID 25681861
- [Background] Francis AM, Haugen CE, Grimes LM, Crow JR, Yi M, Mittendorf EA, Bedrosian I, Caudle AS, Babiera GV, Krishnamurthy S, Kuerer HM, Hunt KK. Is Sentinel Lymph Node Dissection Warranted for Patients with a Diagnosis of Ductal Carcinoma In Situ? Ann Surg Oncol. 2015 Dec;22(13):4270-9. doi: 10.1245/s10434-015-4547-7. Epub 2015 Apr 24. PMID 25905585
- [Background] Julian TB, Land SR, Fourchotte V, Haile SR, Fisher ER, Mamounas EP, Costantino JP, Wolmark N. Is sentinel node biopsy necessary in conservatively treated DCIS? Ann Surg Oncol. 2007 Aug;14(8):2202-8. doi: 10.1245/s10434-007-9353-4. Epub 2007 May 30. PMID 17534687
- [Background] Cox CE, Nguyen K, Gray RJ, Salud C, Ku NN, Dupont E, Hutson L, Peltz E, Whitehead G, Reintgen D, Cantor A. Importance of lymphatic mapping in ductal carcinoma in situ (DCIS): why map DCIS? Am Surg. 2001 Jun;67(6):513-9; discussion 519-21. PMID 11409797
- [Background] Klauber-DeMore N, Tan LK, Liberman L, Kaptain S, Fey J, Borgen P, Heerdt A, Montgomery L, Paglia M, Petrek JA, Cody HS, Van Zee KJ. Sentinel lymph node biopsy: is it indicated in patients with high-risk ductal carcinoma-in-situ and ductal carcinoma-in-situ with microinvasion? Ann Surg Oncol. 2000 Oct;7(9):636-42. doi: 10.1007/s10434-000-0636-2. PMID 11034239
- [Background] Schmale I, Liu S, Rayhanabad J, Russell CA, Sener SF. Ductal carcinoma in situ (DCIS) of the breast: perspectives on biology and controversies in current management. J Surg Oncol. 2012 Feb;105(2):212-20. doi: 10.1002/jso.22020. Epub 2011 Jul 12. PMID 21751217
- [Background] Archer S, Winchester DS. Noninvasive breast cancer. In: Berger DH, Feig BW, Fuhrman GM, eds. The M.D.Anderson Surgical Oncology Handbook. Boston, Mass: Little Brown & Co; 1995:1-11.
- [Background] Shapiro-Wright HM, Julian TB. Sentinel lymph node biopsy and management of the axilla in ductal carcinoma in situ. J Natl Cancer Inst Monogr. 2010;2010(41):145-9. doi: 10.1093/jncimonographs/lgq026. PMID 20956820
- [Background] Fisher B. Role of science in the treatment of breast cancer when tumor multicentricity is present. J Natl Cancer Inst. 2011 Sep 7;103(17):1292-8. doi: 10.1093/jnci/djr240. Epub 2011 Jul 15. PMID 21765010
- [Background] Virnig BA, Shamliyan T, Tuttle TM, Kane RL, Wilt TJ. Diagnosis and management of ductal carcinoma in situ (DCIS). Evid Rep Technol Assess (Full Rep). 2009 Sep;(185):1-549. PMID 20629475
- [Background] SEER. Attachment A for the SEER-MEDICARE PEDSF File. Available at http://healthcaredelivery.cancer.gov/seermedicare/aboutdata/pedsf_attachment_a.pdf. Accessed on March 18, 2016.
- [Background] D'Agostino RB Jr. Propensity score methods for bias reduction in the comparison of a treatment to a non-randomized control group. Stat Med. 1998 Oct 15;17(19):2265-81. doi: 10.1002/(sici)1097-0258(19981015)17:193.0.co;2-b. PMID 9802183
- [Background] Yu JB, Soulos PR, Herrin J, Cramer LD, Potosky AL, Roberts KB, Gross CP. Proton versus intensity-modulated radiotherapy for prostate cancer: patterns of care and early toxicity. J Natl Cancer Inst. 2013 Jan 2;105(1):25-32. doi: 10.1093/jnci/djs463. Epub 2012 Dec 14. PMID 23243199
- [Background] Austin PC. Statistical criteria for selecting the optimal number of untreated subjects matched to each treated subject when using many-to-one matching on the propensity score. Am J Epidemiol. 2010 Nov 1;172(9):1092-7. doi: 10.1093/aje/kwq224. Epub 2010 Aug 28. PMID 20802241
- [Background] Agresti A, Min Y. Effects and non-effects of paired identical observations in comparing proportions with binary matched-pairs data. Stat Med. 2004 Jan 15;23(1):65-75. doi: 10.1002/sim.1589. PMID 14695640
- [Background] Austin PC. The performance of different propensity-score methods for estimating relative risks. J Clin Epidemiol. 2008 Jun;61(6):537-45. doi: 10.1016/j.jclinepi.2007.07.011. Epub 2008 Feb 14. PMID 18471657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because this study is 1) secondary data analysis of an existing database, 2) has two aims using the most recent data when conducting the analyses, and 3) uses Mehalanobis matching, the number of participants in Enrollment is the number of patients who are eligible to our inclusion criteria.
Groups:
- Aim 1 Cohort - SLNB: The Aim 1 Cohort is constructed to perform analysis to address study objective Aim 1. The cohort population include patients older than 67 years old who have received BCS as their first surgery. The time period for defining the cohort is between January 1998 and December 2011. Patients in this group received SLNB.
  Sentinel lymph node biopsy (SLNB): Intervention is defined as that the DCIS patient has undergone SLNB. Patients in each cohort (group) include those who underwent SLNB (intervention) and those who did not (control).
- Aim 1 Cohort - No SLNB: The Aim 1 Cohort is constructed to perform analysis to address study objective Aim 1. The cohort population include patients older than 67 years old who have received BCS as their first surgery. The time period for defining the cohort is between January 1998 and December 2011. Patients in this group did not receive SLNB.
  Sentinel lymph node biopsy (SLNB): Intervention is defined as that the DCIS patient has undergone SLNB. Patients in each cohort (group) include those who underwent SLNB (intervention) and those who did not (control).
- Aim 2 Cohort - SLNB: The Aim 2 Cohort is constructed to perform analysis to address study objective Aim 2.The cohort population include patients older than 67 years old who have received BCS as the final treatment for their DCIS. The time period for defining the cohort is between January 2001 and December 2013. Patients in this group received sentinel lymph node biopsy (SLNB).
  Sentinel lymph node biopsy (SLNB): Intervention is defined as that the DCIS patient has undergone SLNB. Patients in each cohort (group) include those who underwent SLNB (intervention) and those who did not (control).
- Aim 2 Cohort - No SLNB: The Aim 2 Cohort is constructed to perform analysis to address study objective Aim 2.The cohort population include patients older than 67 years old who have received BCS as the final treatment for their DCIS. The time period for defining the cohort is between January 2001 and December 2013. Patients in this group did not receive sentinel lymph node biopsy (SLNB).
  Sentinel lymph node biopsy (SLNB): Intervention is defined as that the DCIS patient has undergone SLNB. Patients in each cohort (group) include those who underwent SLNB (intervention) and those who did not (control).
Period: Overall Study
Arm/Group | Aim 1 Cohort - SLNB | Aim 1 Cohort - No SLNB | Aim 2 Cohort - SLNB | Aim 2 Cohort - No SLNB
Started | 2409 (The sample prior to Mahalanobis matching.) | 13106 (The sample prior to Mahalanobis matching.) | 1992 (The sample prior to Mahalanobis matching.) | 10784 (The sample prior to Mahalanobis matching.)
Completed | 2409 (The sample after Mahalanobis matching; that is, the number in the main analyses.) | 4718 (The sample after Mahalanobis matching; that is, the number in the main analyses.) | 1992 (The sample after Mahalanobis matching; that is, the number in the main analyses.) | 3965 (The sample after Mahalanobis matching; that is, the number in the main analyses.)
Not Completed | 0 | 8388 | 0 | 6819

BASELINE CHARACTERISTICS:
Population: Mahalanobis matching was used to adjust for baseline characteristics and account for potential treatment bias, where those who receive sentinel lymph node biopsy (SLNB) might be systematically different from those who do not. The final matched Aim 1 & 2 cohorts were used for analyses.
Groups:
- Aim 1 Cohort: No SLNB: The Aim 1 Cohort is constructed to perform analysis to address study objective Aim 1. The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 1998 and December 2011, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who did not receive sentinel lymph node biopsy (SLNB) were included (control group).
- Aim 1 Cohort: SLNB: The Aim 1 Cohort is constructed to perform analysis to address study objective Aim 1. The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 1998 and December 2011, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who received sentinel lymph node biopsy (SLNB) were included (intervention group).
- Aim 2 Cohort: No SLNB: The Aim 2 Cohort is constructed to perform analysis to address study objective Aim 2.The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 2001 and December 2013, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who did not receive sentinel lymph node biopsy (SLNB) were included (control group).
- Aim 2 Cohort: SLNB: The Aim 2 Cohort is constructed to perform analysis to address study objective Aim 2.The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 2001 and December 2013, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who received sentinel lymph node biopsy (SLNB) were included (intervention group).
- Total: Total of all reporting groups
Arm/Group | Aim 1 Cohort: No SLNB | Aim 1 Cohort: SLNB | Aim 2 Cohort: No SLNB | Aim 2 Cohort: SLNB | Total
Number analyzed (Participants) | 4718 | 2409 | 3965 | 1992 | 13084
Age, Customized [Count of Participants; unit: Participants]
  67-69 years old | 981 | 573 | 808 | 478 | 2840
  70-74 years old | 1592 | 783 | 1309 | 651 | 4335
  75-79 years old | 1263 | 614 | 1110 | 503 | 3490
  80-84 years old | 670 | 333 | 567 | 272 | 1842
  85+ years old | 212 | 106 | 171 | 88 | 577
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4718 | 2409 | 3965 | 1992 | 13084
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 221 | 135 | 190 | 106 | 652
  Not Hispanic or Latino | 4497 | 2274 | 3775 | 1886 | 12432
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4099 | 2148 | 3494 | 1778 | 11519
  Black | 386 | 170 | 271 | 129 | 956
  Other | 233 | 91 | 200 | 85 | 609
Region of Enrollment [Number; unit: participants]
  United States | 4718 | 2409 | 3965 | 1992 | 13084
Marital Status [Count of Participants; unit: Participants]
  Married | 2286 | 1227 | 1977 | 1038 | 6528
  Unmarried | 2196 | 1085 | 1798 | 867 | 5946
  Other | 236 | 97 | 190 | 87 | 610
Tumor Grade [Count of Participants; unit: Participants]
  Well differentiated | 498 | 254 | 424 | 207 | 1383
  Moderately differentiated | 1371 | 629 | 1278 | 536 | 3814
  Poorly differentiated | 1449 | 802 | 1262 | 730 | 4243
  Undifferentiated | 601 | 321 | 434 | 226 | 1582
  Unknown | 799 | 403 | 567 | 293 | 2062
Tumor size [Count of Participants; unit: Participants]
  <2.0 cm | 2552 | 1264 | 2407 | 1148 | 7371
  2.0-<5.0 cm | 749 | 434 | 550 | 347 | 2080
  >5.0 cm | 149 | 89 | 80 | 42 | 360
  Missing | 1268 | 622 | 928 | 455 | 3273
Hormone receptors [Count of Participants; unit: Participants]
  ER- and PR- | 631 | 341 | 485 | 284 | 1741
  ER+ and PR+ | 2608 | 1329 | 2316 | 1170 | 7423
  Missing | 1479 | 739 | 1164 | 538 | 3920
Comedonecrosis [Count of Participants; unit: Participants]
  Yes | 524 | 297 | 428 | 259 | 1508
  No | 4194 | 2112 | 3537 | 1733 | 11576
Surgeon Volume [Count of Participants; unit: Participants] — "Surgeon volume" reflects women who saw a provider who performed breast conserving surgery on a certain number of women in our sample for the year of this woman's surgery. The larger the number, the larger the provider's patient volume.
  Participants
    1 | 2182 | 1140 | 1986 | 945 | 6253
    2 | 1099 | 578 | 969 | 496 | 3142
    3 | 596 | 329 | 465 | 267 | 1657
    4+ | 727 | 300 | 509 | 266 | 1802
    Not assigned | 114 | 62 | 36 | 18 | 230
Elixhauser Comorbidity [Count of Participants; unit: Participants] — Elixhauser comorbidity measure: 0 (no comorbidity) to 30 (multiple comorbidities), is a claim-based comorbidity index, that requires the diagnosis code to appear on either an inpatient claim or >= 2 outpatient claims greater than 30 days apart in order for the condition to be considered present.
  Participants
    None | 2229 | 1219 | 1955 | 980 | 6383
    1 to 2 | 1914 | 935 | 1548 | 780 | 5177
    3 or more | 575 | 255 | 462 | 232 | 1524
Year of Diagnosis [Count of Participants; unit: Participants]
  1998-1999 | 63 | 30 | 0 | 0 | 93
  2000-2003 | 806 | 395 | 605 | 240 | 2046
  2004-2005 | 863 | 431 | 531 | 264 | 2089
  2006-2007 | 986 | 508 | 647 | 329 | 2470
  2008-2009 | 1048 | 539 | 713 | 380 | 2680
  2010-2011 | 952 | 506 | 753 | 395 | 2606
  2012-2013 | 0 | 0 | 716 | 384 | 1100
Geographic Region [Count of Participants; unit: Participants]
  Midwest | 583 | 296 | 460 | 229 | 1568
  Northeast | 979 | 488 | 763 | 378 | 2608
  South | 1141 | 588 | 1026 | 522 | 3277
  West | 2015 | 1037 | 1716 | 863 | 5631

OUTCOME MEASURES:

1. Primary Outcome: Side Effects (Claim-based Measure), Including Lymphedema, Seroma, Wound Infection, or Pain
Description: Primary outcomes for Aim 1: Acute and subacute side effects include any complication, lymphedema, seroma, wound infection, and pain.
Time Frame: From the first BCS to 9 months post-diagnosis.
Population: Mahalanobis matching was used to adjust for baseline characteristics to account for potential treatment selection bias, where those who received SLNB might be systematically different from those who did not. Matches were assigned by choosing the two best non-SLNB patient matches for each SLNB patient. The final matched cohort was used for analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Matched Aim 1 Cohort: No SLNB: The Aim 1 Cohort was constructed to perform analysis to address study objective Aim 1. The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 1998 and December 2011, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who did not receive sentinel lymph node biopsy (SLNB) were included (control group).
- Matched Aim 1 Cohort: SLNB: The Aim 1 Cohort was constructed to perform analysis to address study objective Aim 1. The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 1998 and December 2011, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who received sentinel lymph node biopsy (SLNB) were included (intervention group).
Arm/Group | Matched Aim 1 Cohort: No SLNB | Matched Aim 1 Cohort: SLNB
Number analyzed (Participants) | 4718 | 2409
Participants
  Number of participants with any side effects | 534 | 404
  Number of participants with lymphedema | 23 | 60
  Number of participants with wound Infection | 453 | 296
  Number of participants with seroma | 179 | 153
  Number of participants with pain | 365 | 237
Statistical Analysis 1: Comparison: Matched Aim 1 Cohort: No SLNB vs Matched Aim 1 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and any complication in the Aim 1 matched cohort; Test type: Other; p < .001, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Odds Ratio (OR) = 1.39, 99% CI 2-sided [1.18 to 1.63] — Reference is no SLNB. Odds ratio accounts for matching and adjusted for subsequent mastectomy within 180 days after initial BCS, prior MRI, and radiation therapy status
Statistical Analysis 2: Comparison: Matched Aim 1 Cohort: No SLNB vs Matched Aim 1 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and lymphedema in the Aim 1 matched cohort; Test type: Other; p < .001, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Odds Ratio (OR) = 4.45, 99% CI 2-sided [2.27 to 8.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Matched Aim 1 Cohort: No SLNB vs Matched Aim 1 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and wound infection in the Aim 1 matched cohort; Test type: Other; p < .001, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Odds Ratio (OR) = 1.24, 99% CI 2-sided [1.00 to 1.54] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Matched Aim 1 Cohort: No SLNB vs Matched Aim 1 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and seroma in the Aim 1 matched cohort; Test type: Other; p < .001, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Odds Ratio (OR) = 1.40, 99% CI 2-sided [1.03 to 1.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Matched Aim 1 Cohort: No SLNB vs Matched Aim 1 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and pain in the Aim 1 matched cohort; Test type: Other; p = .003, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Odds Ratio (OR) = 1.31, 99% CI 2-sided [1.04 to 1.65] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Receipt of Mastectomy
Description: Secondary outcomes for Aim 1: receipt of mastectomy with and without SLNB after initial BCS through 6 months after DCIS diagnosis.
Time Frame: 6 months within DCIS diagnosis
Population: Mahalanobis matching was used to adjust for baseline characteristics and account for potential treatment selection bias, where those who receive SLNB might be systematically different from those who do not. Matches were assigned by choosing the two best non-SLNB patient matches for each SLNB patient. The final matched sample was used for analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Matched Aim 1 Cohort: No SLNB: The Aim 1 Cohort is constructed to perform analysis to address study objective Aim 1. The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 1998 and December 2011, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who did not receive sentinel lymph node biopsy (SLNB) were included (control group).
- Matched Aim 1 Cohort: SLNB: The Aim 1 Cohort is constructed to perform analysis to address study objective Aim 1. The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 1998 and December 2011, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who received sentinel lymph node biopsy (SLNB) were included (intervention group).
Arm/Group | Matched Aim 1 Cohort: No SLNB | Matched Aim 1 Cohort: SLNB
Number analyzed (Participants) | 4718 | 2409
Participants
  Yes | 237 | 413
  No | 4481 | 1996
Statistical Analysis 1: Comparison: Matched Aim 1 Cohort: No SLNB vs Matched Aim 1 Cohort: SLNB; Testing the association between receipt of SLNB and receipt of mastectomy within 6 months of DCIS diagnosis; Test type: Other; p < .001, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01

3. Secondary Outcome: Receipt of Radiation Therapy
Description: Secondary outcomes for Aim 1: Receipt of radiation therapy within 9 months of DCIS diagnosis.
Time Frame: 9 months within DCIS diagnosis
Population: Mahalanobis matching was used to adjust for baseline characteristics and account for potential treatment selection bias, where those who receive SLNB might be systematically different from those who do not. Matches were assigned by choosing the two best non-SLNB patient matches for each SLNB patient. The final matched cohort was used for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Aim 1 Cohort: No SLNB | Matched Aim 1 Cohort: SLNB
Number analyzed (Participants) | 4718 | 2409
Participants
  Yes | 2814 | 1416
  No | 1904 | 993
Statistical Analysis 1: Comparison: Matched Aim 1 Cohort: No SLNB vs Matched Aim 1 Cohort: SLNB; Testing the association between receipt of SLNB and receipt of radiation therapy within 9 months of DCIS diagnosis; Test type: Other; p = .48, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01

4. Secondary Outcome: Overall Survival
Description: Secondary outcomes for Aim 2.
Time Frame: From 9 months post-diagnosis to death/end of study period (up to 1.5 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Matched Aim 2 Cohort: No SLNB: The Aim 2 Cohort is constructed to perform analysis to address study objective Aim 2.The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 2001 and December 2013, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who did not receive sentinel lymph node biopsy (SLNB) were included (control group).
- Matched Aim 2 Cohort: SLNB: The Aim 2 Cohort is constructed to perform analysis to address study objective Aim 2.The cohort population includes patients diagnosed at age 67-94 years with DCIS between January 2001 and December 2013, and had received BCS as their first surgery within 6 months of diagnosis.
  Only those who received sentinel lymph node biopsy (SLNB) were included (intervention group).
Arm/Group | Matched Aim 2 Cohort: No SLNB | Matched Aim 2 Cohort: SLNB
Number analyzed (Participants) | 3965 | 1992
Participants | 727 | 287
Statistical Analysis 1: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and overall mortality in the Aim 2 matched cohort; Test type: Other; p < .001, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 0.88, 99% CI 2-sided [0.73 to 1.05] — Reference is no SLNB. Estimates are from matched cohort and adjusted for physician visits, any hospitalization in the 3-24 months prior to DCIS diagnosis, use of preoperative breast MRI, surgeon's operation volume, and receipt of radiation therapy

5. Secondary Outcome: Lasting Side Effects (Claim-based Measure), Including Lymphedema, Seroma, Wound Infection, or Pain
Description: Secondary outcomes for Aim 2: unadjusted side effects (any side effects, lymphedema, any infection, seroma, pain) in the matched sample by use of sentinel lymph node biopsy (SLNB). Any side effects refer to the occurrence of one or more of the following complications since diagnosis of DCIS: lymphedema related complications, any infection, seroma, and any pain.
Time Frame: From 9 months post-diagnosis to death/end of study period (up to 1.5 years)
Population: Mahalanobis matching was used to adjust for baseline characteristics and account for potential treatment selection bias, where those who receive SLNB might be systematically different from those who do not. Matches were assigned by choosing the two best non-SLNB patient matches for each patient. The final matched cohort was used for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Aim 2 Cohort: No SLNB | Matched Aim 2 Cohort: SLNB
Number analyzed (Participants) | 3965 | 1992
Participants
  Number of participants with any side effects | 2329 | 1204
  Number of participants with lymphedema | 159 | 123
  Number of participants with any infection | 1579 | 751
  Number of participants with seroma | 294 | 186
  Number of participants with pain | 1283 | 701
Statistical Analysis 1: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and any side effects in the matched Aim 2 cohort; Test type: Other; p = 0.207, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 1.09, 99% CI 2-sided [1.00 to 1.20] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and lymphedema related complications in the Aim 2 matched cohort; Test type: Other; p < .001, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 1.53, 99% CI 2-sided [1.12 to 2.11] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and any infection in the Aim 2 matched cohort; Test type: Other; p = 0.113, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 0.98, 99% CI 2-sided [0.87 to 1.10] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and seroma in the Aim 2 matched cohort; Test type: Other; p = 0.010, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 1.21, 99% CI 2-sided [0.93 to 1.58] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and pain in the Aim 2 matched cohort; Test type: Other; p = 0.029, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 1.10, 99% CI 2-sided [0.98 to 1.25] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Breast Cancer Specific Mortality
Description: Primary outcomes for Aim 2: Breast cancer specific mortality from 9 months post-diagnosis to death or the end of the study period (December, 2014).
Time Frame: From 9 months post-diagnosis to death/end of study period (up to 1.5 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Aim 2 Cohort: No SLNB | Matched Aim 2 Cohort: SLNB
Number analyzed (Participants) | 3965 | 1992
Participants | 36 | 19
Statistical Analysis 1: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between between use of sentinel lymph node biopsy (SLNB) and breast cancer specific mortality; Test type: Other; p = 0.861, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 1.13, 99% CI 2-sided [0.54 to 2.35] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Ipsilateral Invasive Breast Cancer Occurrence
Description: Primary outcomes for Aim 2: Ipsilateral invasive breast cancer occurrence after 9 months of a DCIS diagnosis, per SEER reports.
Time Frame: From 9 months post-diagnosis to death/end of study period (up to 1.5 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Aim 2 Cohort: No SLNB | Matched Aim 2 Cohort: SLNB
Number analyzed (Participants) | 3965 | 1992
Participants | 150 | 70
Statistical Analysis 1: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and ipsilateral invasive breast cancer occurrence for the Aim 2 matched cohort; Test type: Other; p = 0.603, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 1.03, 99% CI 2-sided [0.71 to 1.51] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Treated Recurrence
Description: Primary outcomes for Aim 2: Treated recurrence was defined by the receipt of mastectomy after 9 months of a DCIS diagnosis in the Aim 2 matched cohort.
Time Frame: From 9 months post-diagnosis to death/end of study period (up to 1.5 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Aim 2 Cohort: No SLNB | Matched Aim 2 Cohort: SLNB
Number analyzed (Participants) | 3965 | 1992
Participants | 145 | 78
Statistical Analysis 1: Comparison: Matched Aim 2 Cohort: No SLNB vs Matched Aim 2 Cohort: SLNB; Testing the association between use of sentinel lymph node biopsy (SLNB) and treated recurrence in the Aim 2 matched cohort; Test type: Other; p = 0.620, Chi-squared — P-value is unadjusted. Threshold for statistical significance is 0.01; Hazard Ratio (HR) = 1.17, 99% CI 2-sided [0.81 to 1.69] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Not applicable: This project involves secondary data analysis of an existing data-set; thus, we did not collect adverse event data.
Description: We do not collect adverse event information.
Groups:
- EG000: As a retrospective data analysis, we do not collect adverse event information.
Arm/Group | EG000
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT02908178/Prot_SAP_000.pdf